CLINICAL TRIAL: NCT07236645
Title: Efficacy and Safety of Ginkgo Biloba Extract EGb761® in Patients With Diabetic Retinopathy: A Single-Center, Open-Label, Parallel-Group Controlled Trial
Brief Title: Efficacy and Safety of Ginkgo Biloba Extract EGb761® in Patients With Diabetic Retinopathy
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Kun Liu, Chief Physician, Professor, Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 20250716102337760
Record Dates: First submitted 2025-10-08; First posted 2025-11-19 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Non-proliferative Diabetic Retinopathy (NPDR)
MeSH Terms: interventions — ginaton; Ginkgo biloba extract

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ginaton (ginkgo biloba extract tablet) (Experimental)
  Interventions: Drug: Ginaton (ginkgo biloba extract tablet); Other: standard treatment
- Control (Other): standard treatment
  Interventions: Other: standard treatment

INTERVENTIONS:
Drug: Ginaton (ginkgo biloba extract tablet) — Patients in the Ginaton arm, in addition to receiving standard treatment, were administered Ginaton orally at a dose of two tablets (40 mg/tablet) three times daily (after morning, noon, and evening meals) for 2 years, starting from enrollment
  Arms: Ginaton (ginkgo biloba extract tablet)
Other: standard treatment — standard treatment

SUMMARY:
This study is a single-center, open-label, parallel-controlled trial, scheduled to commence in October 2025 at the outpatient and inpatient departments of Shanghai General Hospital. Eligible patients with diabetes mellitus and/or non-proliferative diabetic retinopathy (NPDR), who meet the inclusion and exclusion criteria, will be recruited. General and disease-related information will be collected. All eligible participants will be required to voluntarily sign an informed consent form after fully understanding and accepting the study. Successfully enrolled subjects will be randomly assigned to the Ginaton group or the conventional treatment group, and will receive the corresponding interventions as specified in the study protocol. Follow-up assessments will include blood pressure, blood glucose, glycated hemoglobin, blood lipids, hemorheological parameters, glomerular filtration rate, microalbuminuria, nerve conduction velocity by electromyography, visual acuity, wide-field fundus photography, quality of life (SF-36 questionnaire), and adverse events. The study aims to evaluate the efficacy and safety of ginkgo biloba extract tablet in preventing the development of diabetic retinopathy in patients with long-standing diabetes, as well as in treating patients with mild to moderate NPDR without concomitant diabetic macular edema (DME).

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18 years or older, regardless of gender;
2. Meeting the diagnostic criteria for diabetes mellitus with glycated hemoglobin (HbA1c) ≤13%;
3. Having a diabetes duration ≥5 years without diagnosed diabetic retinopathy or, according to the DR staging criteria proposed by the Group of Fundus Diseases, Ophthalmology Society of Chinese Medical Association in 2014, having at least one eye diagnosed with Stage I or II non-proliferative diabetic retinopathy (NPDR) without concomitant diabetic macular edema (DME);
4. Voluntarily signing the informed consent form.

Exclusion Criteria:

1. Pregnant or lactating women.
2. Poorly controlled hypertension (defined as ≥180/100 mmHg).
3. Patients with coexisting ocular pathologies, such as glaucoma or cataract.
4. Patients with severe impairment of cardiac, pulmonary, hepatic, or renal function, or coagulation disorders, e.g., alanine aminotransferase (ALT) ≥2 times the upper limit of normal (ULN), aspartate aminotransferase (AST) ≥2 ULN, total bilirubin (BIL) ≥1.5 ULN, or estimated glomerular filtration rate (eGFR) ≤30 mL/min/1.73 m².
5. Patients with comorbid psychiatric or neurological disorders.
6. Patients with a known allergy to any component of the investigational product.
7. Patients who received Ginkgo biloba extract treatment within the past 12 months.
8. Patients with a history of intraocular treatments, such as panretinal photocoagulation (PRP), and/or anti-vascular endothelial growth factor (VEGF) therapy, and/or ocular surgery.
9. Patients with a history of cardiovascular events or conditions requiring long-term anticoagulation therapy, such as deep vein thrombosis, pulmonary embolism, atrial fibrillation, or cardiac valve replacement.
10. Any contraindication that, in the investigator's judgment, could limit clinical assessment or treatment.
11. Concurrent participation in any other clinical trial.
12. Patients deemed by the investigator to be unsuitable for inclusion in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-11-20 (Estimated); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Retinal Vessel Density | 2 years
  The difference between groups in the change of retinal vessel density from baseline within 2 years of treatment (at month 24), assessed by OCTA.
Vessel Length Density | 2 years
  The difference between groups in the change of vessel length density from baseline within 2 years of treatment (at month 24), assessed by OCTA.
Vascular Index | 2 years
  The difference between groups in the change of vascular index from baseline within 2 years of treatment (at month 24), assessed by OCTA.
Perfusion Area | 2 years
  The difference between groups in the change of perfusion area from baseline within 2 years of treatment (at month 24), assessed by OCTA.
Choroidal Vessel Volume | 2 years
  The difference between groups in the change of choroidal vessel volume from baseline within 2 years of treatment (at month 24), assessed by OCTA.
Foveal Avascular Zone Area | 2 years
  The difference between groups in the change of foveal avascular zone area from baseline within 2 years of treatment (at month 24), assessed by OCTA.
Stromal Volume | 2 years
  The difference between groups in the change of stromal volume from baseline within 2 years of treatment (at month 24), assessed by OCTA.
Stromal Index | 2 years
  The difference between groups in the change of stromal index from baseline within 2 years of treatment (at month 24), assessed by OCTA.

SECONDARY OUTCOMES:
The percentage of glycated hemoglobin (HbA1c) | 2 years
  Differences in the percentage of glycated hemoglobin (HbA1c) between the two groups over the 2-year treatment period.
Urinary Albumin-to-creatinine Ratio （UACR） | 2 years
  Between-group difference in urinary albumin-to-creatinine ratio (UACR) during the 2-year treatment period.
Estimated Glomerular Filtration Rate （eGFR） | 2 years
  Between-group difference in urinary estimated glomerular filtration rate （eGFR） during the 2-year treatment period.
Motor Nerve Conduction Velocity (MNCV) | 2 years
  Differences in motor nerve conduction velocity (MNCV) of the median and common peroneal nerves from baseline at each visit over the 2-year treatment period.
Diabetic Retinopathy Severity Scale (DRSS) score | 2 years
  Baseline ETDRS DRSS: None (level 10); Mild to moderate nonproliferative DR (levels 14, 15, 20, 35, and 43); Moderately severe/severe nonproliferative DR (levels 47 and 53); Mild/moderate/high-risk/advanced proliferative DR (levels 61, 65, 71,75, 81, and 85)
36-item Short-Form (SF-36) score over the 2-year treatment period | 2 years
  Differences in quality of life scores based on the 36-Item Short Form Health Survey between the two groups over the 2-year treatment period.The score for each of the eight health domains and the two summary measures ranges from 0 to 100.A higher score indicates a more favorable health state.
Whole Blood Viscosity | 2 years
  The between-group difference in whole blood viscosity (a hemorheological parameter) during the 2-year treatment period.
Plasma Viscosity | 2 years
  The between-group difference in plasma viscosity (a hemorheological parameter) during the 2-year treatment period.
Hematocrit | 2 years
  The between-group difference in hematocrit (a hemorheological parameter) during the 2-year treatment period.
Fibrinogen | 2 years
  The between-group difference in fibrinogen (a hemorheological parameter) during the 2-year treatment period.
Sensory Nerve Conduction Velocity (SNCV) | 2 years
  Differences in sensory nerve conduction velocity (SNCV) of the median and superficial peroneal nerves from baseline at each visit over the 2-year treatment period.